CLINICAL TRIAL: NCT03852420
Title: Safety and Effectiveness Evaluation of Boston Scientific's Single Shot LUMINIZE RF Balloon Catheter in the Treatment of Symptomatic, Drug Refractory Paroxysmal Atrial Fibrillation
Brief Title: Boston Scientific's Single Shot LUMINIZE RF Balloon Catheter in the Treatment of Symptomatic, Drug Refractory Paroxysmal Atrial Fibrillation
Acronym: VISUALISE AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor discretion
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA002
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The LUMINIZE RF Balloon Catheter is a multi-electrode, irrigated, over-the-wire balloon catheter designed to facilitate cardiac electrophysiological mapping and ablation. The catheter interfaces with the LUMINIZE Console and is designed to localize potentials and create lesions using multi-polar RF energy.
  The System consists of the following devices and components:
  * LUMINIZE RF Balloon Catheter
  * LUMINIZE Steerable Sheath
  * LUMINIZE Console
  * LUMINIZE System Accessories
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment with the LUMINIZE RF Balloon Catheter (Experimental): Subjects undergoing cardiac ablation procedure LUMINIZE™ RF Balloon Catheter System.
  Interventions: Device: LUMINIZE RF Balloon Catheter

INTERVENTIONS:
Device: LUMINIZE RF Balloon Catheter — Ablation Therapy with the LUMINIZE RF Balloon Catheter

SUMMARY:
To establish the safety and effectiveness of the LUMINIZE RF Balloon Catheter System for treatment of symptomatic, drug refractory, recurrent, paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
The VISUALISE AF study is a multi-center (global), open label, prospective, single arm study to establish the safety and effectiveness of the LUMINIZE RF Balloon Catheter System. The planned indication for use within the United States for LUMINIZE RF Balloon Catheter System is for the treatment of drug refractory, recurrent, symptomatic, Paroxysmal Atrial Fibrillation (PAF).

All subjects fitting the enrollment criteria, signing the consent and undergoing the index procedure with the study devices will be followed up for one year.

ELIGIBILITY:
Inclusion Criteria:

1. History of recurrent symptomatic paroxysmal atrial fibrillation (PAF), defined as atrial fibrillation that terminates spontaneously or with intervention (either procedure or drug therapy) within seven days of onset. Minimum documentation includes the following:

   i) a physician's note indicating recurrent self-terminating atrial fibrillation (AF) which includes at least two symptomatic AF episodes documented by patient history within last six months from enrollment, and ii) one electrocardiographically documented AF episode within 12 months prior to enrollment.
2. Subjects who are eligible for an ablation procedure for PAF according to 2017 HRS expert consensus statement on catheter ablation of atrial fibrillation.
3. Subjects refractory or intolerant to at least one class I or III antiarrhythmic medication.
4. Subjects who are willing and capable of providing informed consent.
5. Subjects who are willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center.
6. Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* 1. Any known contraindication to an AF ablation or anticoagulation 2. Continuous AF lasting longer than seven (7) days from onset 3. History of previous left atrial ablation or surgical treatment for AF/AFL/AT 4. Amiodarone use within 90 days prior to enrollment 5. Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause 6. Age>80 years 7. Structural heart disease, heart conditions or implanted devices as described below:

  1. Left ventricular ejection fraction < 40% based on the most recent transthoracic echocardiogram (TTE) performed (≤ 180 days prior to enrollment)+
  2. Left atrial diameter greater than 5.5cm or left atrial volume >50 ml/m² ml indexed based on the most recent TTE performed ≤ 180 days prior to enrollment+
  3. An implanted pacemaker, ICD, CRT device or an arrhythmia loop recorder
  4. Subjects with heart failure and New York Heart Association (NYHA) Class III or IV (≤ 180 days prior to enrollment)
  5. Previous cardiac surgery i.e. ventriculotomy or atriotomy, excluding atriotomy for coronary artery bypass graft (CABG)
  6. Previous cardiac valvular surgical or percutaneous procedure, or prosthetic valve, including mitral valve clips
  7. Interatrial baffle, closure device, patch, or patent foramen ovale (PFO) occluder
  8. Presence of left atrial appendage occlusion device
  9. Presence of any pulmonary vein stents
  10. Documented or suspected stenosis of any pulmonary veins
  11. CABG, percutaneous transluminal coronary angioplasty (PTCA)/ percutaneous coronary intervention (PCI)/ coronary stent procedures within 90 days prior to enrollment
  12. Unstable angina or ongoing myocardial ischemia
  13. Previous myocardial infarction within 90 days prior to enrollment
  14. Moderate or severe mitral stenosis assessed on the most recent TTE ≤180 days prior to enrollment as pulmonary artery systolic pressure >30 mmHg(1)
  15. Vena cava embolic protection filter devices and/ or known femoral thrombus who require catheter insertion from the femoral approach
  16. Evidence of myxoma, left atrial thrombus or intracardiac mural thrombus++ 8. Stage 3B renal disease or higher (estimated glomerular filtration rate, eGFR <45 mL/min) 9. History of blood clotting or bleeding disease 10. Any prior history of documented cerebral infarct, TIA or systemic embolism [excluding a post-operative deep vein thrombosis (DVT)] ≤180 days prior to enrollment 11. Active systemic infection 12. Pregnant, lactating (current or anticipated during study follow up), or women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion) 13. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the sponsor to determine eligibility.

      14. Subjects who in the judgment of the investigator have a life expectancy of less than two years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety event free rate at 12 months post procedure. | 0-12 months post procedure
  Primary safety events will consist of a composite of procedure-related and/or device-related adverse events.
Failure free rate at 12 months post procedure. | 0-12 months post procedure
  Failure defined as:
  * Failure to achieve acute procedural success
  * Use of amiodarone post index procedure
  * Surgical treatment for AF/ AFL/ AT post index procedure
  * Use of a non-study ablation catheter for any AF targets in the index procedure or repeat procedure during the blanking period
  * More than one repeat procedure with the LUMINIZE RF Balloon Catheter during the blanking period
  * Documented atrial fibrillation, or new onset of AFL or AT between days 91 post index procedure and 365 days post index procedure captured by one of the following methods:
  * ≥ 30 seconds in duration from the study specific event monitor or Holter Monitor
  * ≥ 10 seconds 12-lead Electrocardiography (ECG)
  * Any of the following interventions for atrial fibrillation, or new onset of atrial flutter or atrial tachycardia between days 91 post index procedure and 365 days:
  * Repeat procedure
  * Cardioversion for AF/AFL/AT
  * Prescribed any antiarrhythmic drug (AAD)*

SECONDARY OUTCOMES:
Secondary Safety Endpoint | 12 months
  Serious Adverse Events (SAE) and Adverse Events (AE) related to the procedure and/or study device through 12 months post Index Procedure.
Acute procedural success | 1 day
  Rate of acute procedural success defined as the achievement of electrical isolation of all pulmonary veins (PVs) by using the LUMINIZE RF Balloon Catheter system.

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Wazni, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No
No requests for study data have been made at this time, however Boston's Scientific's policy on data sharing can be found at http://www.bostonscientific.com/en-US/data-sharing-requests.html